CLINICAL TRIAL: NCT00235781
Title: Non-Phased Study of the Use of a Single Dose of Thymoglobulin for Immunosuppressive Induction in Renal Transplant Recipients as Compared to a Standard Four Dose Regimen
Brief Title: Single Dose Thymoglobulin for Induction in Adult Renal Allograft Recipients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-0783
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2006-10-16 (Estimated); Status verified 2006-10

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Antilymphocyte Serum; Induction; Graft Rejection
MeSH Terms: interventions — thymoglobulin

INTERVENTIONS:
Drug: Thymoglobulin

SUMMARY:
The aim of this trial is to compare the safety and efficacy of a single dose of Thymoglobulin, rabbit derived antithymocyte globulin (Thymoglobulin, SangStat, Fremont, CA) to our standard four dose, four day Thymoglobulin induction regimen from the time of transplantation through a six month follow-up period. The primary endpoint will be the incidence of acute rejection. Secondary endpoints will include serious adverse events, evaluation of renal function, patient and graft survival, incidence of infectious complications, incidence of post-transplantation lymphoproliferative disorder (PTLD), duration and extent of lymphocyte depletion and immunoassays for evidence of recipient immune response to the allograft as well as duration of hospital stay.

DETAILED DESCRIPTION:
Induction therapy, using polyclonal or monoclonal antibody preparations as an adjunct immunosuppressive agent during the initial transplant period, has helped to decrease the incidence of acute rejection significantly. In the 1980's acute rejection occurred in approximately 50% of renal transplant recipients. In the current era of transplantation, the combination of potent induction agents and newly available maintenance immunosuppressive agents has reduced the acute rejection rate to less than 20% at most transplant centers. Our center has routinely achieved acute rejection rates of approximately 5% using a standard induction protocol with the polyclonal antibody agent Thymoglobulin.

Preventing acute rejection significantly decreases the requirement for re-hospitalization, the need for diagnostic renal allograft biopsy and subsequent exposure to high dose corticosteroids and other immunosuppressive agents. The threat of early allograft loss secondary to rejection refractory to treatment or permanent injury and shortened graft survival following treatment of a severe rejection is also circumvented.

Polyclonal antibody preparations are produced by immunizing animals with human lymphocytes or thymocytes. Polyclonal antibody preparations are approved for treatment of acute renal allograft rejection, but are routinely used as induction agents and for prevention of rejection in all solid organ allografts. Commercially available preparations in the United States are equine/thymocyte derived (Atgam, Pharmacia & Upjohn, Kalamazoo, MI) and rabbit/thymocyte derived (Thymoglobulin, Genzyme, Cambridge, MA).

Rabbit derived preparations are thought to be potentially more efficacious than equine derived products. Studies performed at this renal transplant center demonstrated that Thymoglobulin has superior efficacy compared to Atgam in the prevention of rejection (1). Not only was the acute rejection rate lower, but graft survival was also better at 1 and 5-years (1). [Hardinger, 2004 #18]. This result has been attributed in part to a more pronounced and prolonged lymphopenia induced by Thymoglobulin (2).

The broad specificity of polyclonal agents to multiple cell signaling and adhesion molecules provides a theoretic advantage compared to monoclonal antibodies. In addition to inducing a profound and prolonged lymphopenia through complement-dependent lysis or by opsonization and phagocytosis, the broad specificity of polyclonal antibody agents affects multiple costimulatory and adhesion molecules involved in cellular and antibody mediated immune processes. The effects on adhesion molecules, cytokines, chemokines and platelets may be critical to the noted decrease in the incidence of delayed renal allograft function associated with initiation of Thymoglobulin therapy intraoperatively (3). Prevention of delayed graft function may also subsequently decrease the incidence of acute rejection and prolong allograft survival.

The use of a potent induction agent such as Thymoglobulin also allows for a delayed introduction of maintenance immunosuppression with calcineurin inhibitors in the immediate post-transplant setting. The ability to delay the introduction of therapeutic doses of calcineurin inhibitors, when necessary, can also assist in decreasing the incidence of delayed graft function and simplifies patient management in this time period.

Thymoglobulin has now become the preferred polyclonal agent used for induction in renal transplantation. The most recent complete yearly data from the Scientific Registry of Transplant Recipients in 2003 indicated that 70% of all renal transplant recipients in that calendar year received some form of induction therapy. Thymoglobulin (34% of patients) was the most commonly administered agent, while one of two available monoclonal antibody preparations directed against the interleukin-2 receptor (IL2-R) was administered to approximately 35% of renal transplant recipients (4).

When Thymoglobulin is used in the treatment of acute rejection, a total dose of 10-12mg/kg is often administered over the course of several days (5). The optimal dose of Thymoglobulin that should be administered for induction is unclear, although a primate model suggests a total human equivalent dose of approximately 6mg/kg may be appropriate (6). Most transplant centers using Thymoglobulin for induction have administered a total dose of 6-10mg/kg, given at varying intervals (usually daily or every other day) with each individual dose usually given as 1 to 1.5mg/kg/day over approximately six hours. Our standard induction protocol has been 1.5mg/kg/day for a total of four doses (total dose 6mg/kg).

The ability to administer Thymoglobulin as a single, large dose has several potential pharmacoeconomic benefits. This administration protocol would simplify post-transplant care in the hospital and allow for earlier patient discharge. Cost savings would result from both a shorter hospital stay and decreased administration costs associated with fewer intravenous administrations.

The administration of a single, large dose infusion of Thymoglobulin has been used in an attempt to induce "prope´" (Latin for almost) allograft tolerance (7). In this study, that included 50 renal allograft recipients, a single dose infusion of Thymoglobulin (5mg/kg) was used in conjunction with a marked minimization of maintenance immunosuppression. The induction protocol was well tolerated, and maintenance immunosuppression consisted of monotherapy with tacrolimus.

Another study described the administration of Thymoglobulin 5mg/kg/day given as two separate doses (10mg/kg total) in 39 renal allograft recipients (8). One dose was administered on the day of transplantation and the subsequent dose on post-transplant day number one. No patients in this study were withdrawn secondary to adverse events and the acute rejection rate was 6% with a patient and graft survival of 95% at a mean follow-up of 14.5 months.

We have previously performed a short course Thymoglobulin induction study using an initial dose of 3mg/kg with subsequent doses of 1.5mg/kg on post-transplant days one and two (9). This regimen was well tolerated and resulted in a low acute rejection rate of 5%, a one year graft survival of 95% and earlier hospital discharge compared to a previously standard seven day Thymoglobulin induction protocol.

Thus, we hypothesize that a single dose of Thymoglobulin (6mg/kg), initiated intraoperatively and administered over the course of 24 hours, will have comparable safety and efficacy as compared to our current standard induction protocol of four separate doses of Thymoglobulin 1.5mg/kg (total dose 6mg/kg). Single dose administration of Thymoglobulin should provide a low rate of acute rejection, a low rate of delayed graft function, allow for delayed introduction of calcineurin inhibitors if indicated, and potentially allow for earlier patient discharge while consuming fewer resources. If this single dose induction protocol demonstrates similar safety and efficacy to our current standard four dose induction protocol, it may become our standard of care. This study may also be a bridge to subsequent dose finding studies for single dose Thymoglobulin administration and subsequent comparative studies of single-dose Thymoglobulin to other induction agents.

1. Brennan DC, Flavin K, Lowell JA, et al. A randomized, double-blinded comparison of Thymoglobulin versus Atgam for induction immunosuppressive therapy in adult renal transplant recipients. Transplantation 1999;67(7):1011-1018.
2. Hardinger KL, Schnitzler MA, Miller B, et al. Five-year follow up of thymoglobulin versus ATGAM induction in adult renal transplantation. Transplantation 2004;78(1):136-141.
3. Goggins WC, Pascual MA, Powelson JA, et al. A prospective, randomized, clinical trial of intraoperative versus postoperative Thymoglobulin in adult cadaveric renal transplant recipients. Transplantation 2003;76(5):798-802.
4. Shapiro R, Young JB, Milford EL, et al. Immunosuppression: evolution in practice and trends, 1993-2003. Am J Transplant 2005;5(4 Pt 2):874-886.
5. Gaber AO, First MR, Tesi RJ, et al. Results of the double-blind, randomized, multicenter, phase III clinical trial of Thymoglobulin versus Atgam in the treatment of acute graft rejection episodes after renal transplantation. Transplantation 1998;66(1):29-37.
6. Preville X, Flacher M, LeMauff B, et al. Mechanisms involved in antithymocyte globulin immunosuppressive activity in a nonhuman primate model. Transplantation 2001;71(3):460-468.
7. Starzl TE, Murase N, Abu-Elmagd K, et al. Tolerogenic immunosuppression for organ transplantation. Lancet 2003;361(9368):1502-1510.
8. Uslu A, Nart A, Coker I, et al. Two-day induction with thymoglobulin in kidney transplantation: risks and benefits. Transplant Proc 2004;36(1):76-79.
9. Agha IA, Rueda J, Alvarez A, et al. Short course induction immunosuppression with thymoglobulin for renal transplant recipients. Transplantation 2002;73(3):473-475.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. All consenting adult renal transplant recipients scheduled to receive induction therapy (deceased donor, living-related, or living-unrelated)
3. Females of childbearing age must have a negative pregnancy test performed at the time of admission for transplantation
4. Patient or guardian agrees to participate in the study and signs the informed consent.
5. No known contraindication to the administration of Thymoglobulin

Exclusion Criteria:

1. A known allergy to rabbit proteins or previous significant intolerance of Thymoglobulin administration
2. Pregnant women or nursing mothers
3. Patients with serological evidence of infection with HIV-1, human T-cell leukemia virus type 1 (HTLV-1), or the presence of serum hepatitis B surface antigen (HBsAg)
4. Recipients of a human leukocyte antigen (HLA) identical living donor renal allograft (2-haplotype match)
5. Recipients of simultaneous multiple organ transplantation
6. Recipients with a pre-existing, non-renal, solid organ transplant
7. Recipients of ≥2 previous renal allografts
8. Patients with a history of malignancy with evidence of recurrence within 2 years (except adequately treated localized squamous or basal cell carcinoma of the skin).
9. Any patient who, in the opinion of the investigator, has a significant medical or psychosocial problem that should preclude them from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2006-01; Study Completion 2006-02

PRIMARY OUTCOMES:
Incidence of acute rejection.

SECONDARY OUTCOMES:
Serious adverse events
renal function
patient and graft survival
infection
PTLD
duration and extent of lymphocyte depletion and immunoassays for evidence of recipient immune response
duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Koch, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States